CLINICAL TRIAL: NCT05388838
Title: Screening for Oculocerebral Lymphoma by Identifying the Phenotype Carried by Circulating NK Cells in Patients with Uveitis
Brief Title: Screening for Oculocerebral Lymphoma with the Phenotype of NK Cells in Patients with Uveitis
Acronym: DeLPHy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL22_0078; 2022-A00254-39 (Other: ANSM)
Record Dates: First submitted 2022-05-16; First posted 2022-05-24 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Uveitis; Lymphoma; NK-Cell Lymphoma
MeSH Terms: conditions — Uveitis; Lymphoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Prospective Case Control Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Negative control (Active Comparator): uveitis patients with a diagnosis other than ocular diagnosis other than ocular lymphoma and without cerebral lymphoma (15 patients),
  Interventions: Biological: Blood sample
- Primary ocular Lymphoma without brain involvementand never treated (Active Comparator): patients with primary ocular lymphoma without brain involvement and never treated (5 patients),
  Interventions: Biological: Blood sample
- Primary ocular Lymphoma without brain involvement and treated (Active Comparator): patients with primary ocular lymphoma without brain involvement, treated and considered in remission (5 patients),
- Primary ocular Lymphoma without brain involvement in relapse (Active Comparator): patients with primary ocular lymphoma without brain involvement, considered in relapse (5 patients),
  Interventions: Biological: Blood sample
- Positive control (Active Comparator): patients with cerebral lymphoma with or without ocular involvement and without uveitis (15 patients).
  Interventions: Biological: Blood sample
- Patients without brain involvement and without uveitis (Active Comparator): Patients presenting for cataract follow-up (pre- or post-operative), glaucoma, retinal detachment or epiretinal membrane, with no brain damage or uveitis (15 patients).
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Blood sample will be taken at D0: 63 ml (7 tubes of 9 ml),
  Arms: Negative control; Patients without brain involvement and without uveitis; Positive control; Primary ocular Lymphoma without brain involvement in relapse; Primary ocular Lymphoma without brain involvementand never treated

SUMMARY:
Uveitis is an inflammation of the uvea, an ocular tunic comprising the iris, ciliary body and choroid. This inflammation can also involve other tissues such as the retina, the optic nerve and the aqueous humor. These diseases can result in significant vision loss and account for 10% of all blindness in developed countries, and up to 25% in developing countries. The main difficulty in this pathology is to make the etiological diagnosis, which then allows a specific treatment of the disease. The main etiologie are inflammatory or infectious (sarcoidosis, tuberculosis) but other cancerous etiologies are possible and are of more complicated diagnosis.

Vitreoretinal lymphoma is a subtype of central nervous system lymphoma, which is generally associated with a poor prognosis. It is a diffuse non-Hodgkin's lymphoma, with large B cells. It can be primary ocular (Primary Intra-Ocular Lymphoma - LIOP), without brain involvement, but can also be secondary to central nervous system involvement, which explains the poor prognosis of the disease. Approximately 50-90% of LIOP develop brain involvement within 1-2 years of diagnosis, which encourages early diagnosis to avoid brain involvement as much as possible.

The main obstacle to rapid diagnosis is the difficulty of identifying LIOP. Indeed, the clinical symptoms of this rare disease are often identical to classical uveitis, and the diagnostic means to detect it are invasive and require a trained ophthalmologist and hematologist team. LIOP diagnostic tests are often delay in the management of uveitis and lead to diagnostic erraticity that can last between 4 to 40 months.

The INSERM U1183 unit is developing a diagnostic technology for lymphomas based on the analysis of blood NK cells and their phenotypes including those acquired by trogocytosis (WO/2016/005548).

A rapid, simple, minimally invasive LIOP test using this technology could therefore be propose to all patients presenting with uveitis and whose clinical criteria could match those of LIOP.

The research hypothesis is : Could the diagnostic wandering of patients with primary intraocular lymphoma be reduced by a rapid blood test for NK cell phenotype of patients with uveitis? Following a simple blood test, a rapid LIOP test, using this diagnostic technology, could therefore be proposed to all patients with uveitis and clinical criteria (age, intermediate and posterior location of the uveitis) corresponding to those of LIOP.

The primary objective of this study is to compare the phenotype of circulating NK cells of patient with untreated intraocular lymphoma versus the phenotype of patient with non-cancerous uveitis.

ELIGIBILITY:
Inclusion Criteria:

GENERAL CRITERIA

* Male or female over 18 years of age,
* Free, informed, written consent signed by the patient and the investigator (at the latest on the day of inclusion) and before any examination required by the research,
* Patient affiliated to the social security system or beneficiary of such a system,
* Maximum volume of sampling (care + research) per 30-day period to be adapted according to the patient's weight (Order of April 12, 2018 establishing the list of research mentioned in 2° of Article L. 1121-1).

SPECIFIC CRITERIA

- Patient affected in one or both eyes: of uveitis with another diagnosis than ocular lymphoma and without cerebral lymphoma (Group 1), or primary ocular lymphoma without brain involvement and never treated (Group 2), or primary ocular lymphoma without brain involvement, treated and considered in remission (IL10 HA level < 10) (Group 3), or primary ocular lymphoma without brain involvement, and considered in relapse (IL10 HA level > 30) (Group 4), or cerebral lymphoma with or without ocular involvement and without uveitis (Group 5), or cataract (pre- and post-op), glaucoma, retinal detachment or epiretinal retinal detachment or epiretinal membrane, but no brain damage or uveitis (group 6).

Exclusion Criteria:

* -GENERAL CRITERIA
* Patient participating in an ongoing clinical trial at the time of the inclusion visit,
* Pregnant women, women in labor or nursing mothers,
* Persons deprived of liberty by a judicial or administrative decision,
* Persons under psychiatric care,
* Persons admitted to a health or social institution for purposes other than research,
* Persons of full age who are subject to a legal protection measure (guardianship, curatorship).

SPECIFIC CRITERIA

* Patient for whom the diagnosis of ocular or cerebral lymphoma is uncertain,
* Patient with another systemic cancer that is evolving or in remission < 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
percentage of NK Cells in blood with phenotype acquired by trogocytosis (WO/2016/005548) in patients with uveitis with a diagnosis other than ocular lymphoma and without cerebral lymphoma (Negative control) | through study completion, an average of 1 year
  mesure by Flow Cytometry
percentage of NK Cells in blood with phenotype acquired by trogocytosis (WO/2016/005548) in patients with primary ocular lymphoma without brain involvement and never treated | through study completion, an average of 1 year
  mesure by Flow Cytometry

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service d'Ophtalmologie, Hôpital de la Croix-Rousse, GHN, Lyon
  - Service d'Hématologie Clinique, Hôpital Lyon Sud, Lyon

IPD SHARING:
Plan to Share IPD: Undecided